CLINICAL TRIAL: NCT00077493
Title: Pediatric Phase I Trial of BL22 for Refractory CD22-Positive Leukemias and Lymphomas
Brief Title: BL22 Immunotoxin In Treating Young Patients With Relapsed or Refractory Acute Lymphoblastic Leukemia or Non-Hodgkin's Lymphoma
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: protocol development and Amended protocol revision
Sponsor: MedImmune LLC (Industry)
Collaborators: Cambridge Antibody Technology (Other)
Responsible Party: Karen Kaucic, M.D., MedImmune Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000352020; NCI-04-C-0079H; NCI-5643; NCT00075309 (obsolete NCT alias)
Record Dates: First submitted 2004-02-10; First posted 2004-02-12 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Leukemia; Lymphoma
Keywords: recurrent childhood acute lymphoblastic leukemia; Burkitt lymphoma; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; childhood non-Hodgkin lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating | interventions — RFB4(dsFv)-PE38 recombinant immunotoxin; Antibodies, Monoclonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): BL22 immunotoxin
  Interventions: Drug: BL22 immunotoxin
- 2 (Active Comparator): antibody therapy
  Interventions: Procedure: antibody-drug conjugate therapy
- 3 (Active Comparator): immunotoxin therapy
  Interventions: Procedure: immunotoxin therapy
- 4 (Active Comparator): monoclonal antibody therapy
  Interventions: Procedure: monoclonal antibody therapy

INTERVENTIONS:
Drug: BL22 immunotoxin — BL22 immunotoxin IV over 30 minutes on days 1, 3, and 5 OR on days 1, 3, 5, 7, 9, and 11. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve a complete response (CR) or unconfirmed CR (CRu) receive 2 additional courses beyond CR or CRu for a maximum of 6 courses.
  Arms: 1
Procedure: antibody-drug conjugate therapy — CD22 antibody, RFB4 on day 7
  Arms: 2
Procedure: immunotoxin therapy — tested for immunogenicity to CAT-8015 before each cycle and at end of study.
  Arms: 3
Procedure: monoclonal antibody therapy — administered intravenously over 30 minutes.
  Arms: 4

SUMMARY:
RATIONALE: BL22 immunotoxin can locate tumor cells and kill them without harming normal cells. BL22 immunotoxin may be effective in treating relapsed or refractory acute lymphoblastic leukemia and non-Hodgkin's lymphoma.

PURPOSE: This phase I trial is studying the side effects and best dose of BL22 immunotoxin in treating young patients with relapsed or refractory acute lymphoblastic leukemia or non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the toxic effects of BL22 immunotoxin in pediatric patients with relapsed or refractory CD22-positive acute lymphoblastic leukemia or non-Hodgkin's lymphoma.
* Determine the maximum tolerated dose of this drug in these patients.
* Determine the immunogenicity of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.

Secondary

* Determine the in vitro cytotoxicity of this drug against lymphoblasts from patients with acute lymphoblastic leukemia.
* Determine the therapeutic efficacy of this drug in inducing remissions in these patients.
* Determine changes in lymphocyte subsets, immunoglobulin levels, serum cytokines, and soluble cytokine receptor levels in patients treated with this drug.

OUTLINE: This is a non-randomized, dose-escalation study.

Patients receive BL22 immunotoxin IV over 30 minutes on days 1, 3, and 5 OR on days 1, 3, 5, 7, 9, and 11. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve a complete response (CR) or unconfirmed CR (CRu) receive 2 additional courses beyond CR or CRu for a maximum of 6 courses.

Cohorts of 3-6 patients receive escalating doses of BL22 immunotoxin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, the cohort is expanded and a total of 12 patients are treated at that dose.

Patients are followed weekly for at least 1 month and then every 1-3 months thereafter.

PROJECTED ACCRUAL: A total of 95 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed acute lymphoblastic leukemia (ALL) or non-Hodgkin's lymphoma (including lymphoblastic lymphoma, Burkitt's lymphoma, and large cell lymphoma)

  * Not amenable to available curative therapies
* Relapsed or refractory disease after at least 1 standard chemotherapy and 1 salvage regimen
* CD22 positive according to at least 1 of the following criteria:

  * More than 15% CD22-positive malignant cells by immunohistochemistry
  * More than 30% CD22-positive malignant cells by fluorescent-activated cell sorter analysis
* Measurable or evaluable disease
* Prior CNS involvement allowed provided there is no current evidence of CNS malignancy
* No CNS leukemia or lymphoma as manifested by any of the following:

  * Cerebrospinal fluid (CSF) WBC ≥ 5/mm^3 and confirmation of CSF blasts
  * Cranial neuropathies secondary to underlying malignancy
  * Radiologically detected CNS lymphoma
* No isolated testicular ALL
* Ineligible for or refused hematopoietic stem cell transplantation OR has disease activity that prohibits the time required to identify a suitable stem cell donor

PATIENT CHARACTERISTICS:

Age

* 6 months to 24 years

Performance status

* ECOG 0-3 (12 to 24 years of age)
* Lansky 40-100% (under 12 years of age)

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics
* Absolute neutrophil count > 1,000/mm^3 *
* Platelet count > 50,000/mm^3 * NOTE: *Non-leukemic patients only

Hepatic

* Bilirubin ≤ 2.0 mg/dL
* AST and ALT ≤ 5 times upper limit of normal
* No active hepatitis B or C infection

Renal

* Creatinine normal for age OR
* Creatinine clearance ≥ 60 mL/min

Immunologic

* No serum neutralization of more than 75% of the activity of 1 µg/mL of study drug
* HIV negative

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No clinically significant unrelated systemic illness that would preclude study participation
* No other significant organ dysfunction that would preclude study participation
* No psychiatric illness or social situation that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* At least 1 week since prior colony-stimulating factors (e.g., filgrastim [G-CSF], sargramostim [GM-CSF], or epoetin alfa)
* Prior autologous or allogeneic hematopoietic stem cell transplantation (HSCT) allowed
* More than 100 days since prior allogeneic HSCT

Chemotherapy

* See Disease Characteristics
* At least 2 weeks since prior chemotherapy (6 weeks for nitrosoureas)

Endocrine therapy

* Concurrent corticosteroids allowed provided there has been no increase in the dose 1 week prior to and after study entry

  * Steroid taper allowed

Radiotherapy

* At least 3 weeks since prior radiotherapy

  * Allowed in the past 3 weeks provided the volume of the bone marrow treated is < 10% AND the patients has measurable disease outside of the radiation port

Surgery

* Not specified

Other

* Recovered from prior therapy
* At least 30 days since prior investigational drugs
* No other concurrent investigational drugs

Ages: 6 Months to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 95 (Estimated)
Dates: Start 2004-01; Primary Completion 2008-10 (Estimated); Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
assessment of efficacy, safety, pharmacokinetics, immunogenicity. | end of study

SECONDARY OUTCOMES:
Expansion of MTD | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Alan S. Wayne, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States